CLINICAL TRIAL: NCT02524678
Title: A Phase I, Placebo-controlled, Randomized, Double Blind, Dose-escalation Study to Assess the Safety and Pharmacokinetic and Pharmacodynamic Characteristics of Repeated-dose URC102 in Healthy Korean Adult Males
Brief Title: Phase 1 Study(Additional) of URC102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URC004KR
Record Dates: First submitted 2015-07-22; First posted 2015-08-17 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — URC102

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- URC102 (Active Comparator): URC102
  Interventions: Drug: URC102

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: URC102
  Arms: URC102

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK and PD of URC102 in healthy subjects.

DETAILED DESCRIPTION:
Tolerability, safety, and pharmacokinetics (PK) of URC102 will be assessed after 7-day repeated oral dose in healthy adult Korean males. In addition, pharmacodynamic (PD) response of blood and urinary uric acid levels will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Participated in other clinical study within past 3 months prior to receiving an IP administration

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2016-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with AE | 2 week

SECONDARY OUTCOMES:
Plasma URC102 concentration | 2 week
Change of plasma uric acid | 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HA, Yu KS, Park SI, Yoon S, Onohara M, Ahn Y, Lee H. URC102, a potent and selective inhibitor of hURAT1, reduced serum uric acid in healthy volunteers. Rheumatology (Oxford). 2019 Nov 1;58(11):1976-1984. doi: 10.1093/rheumatology/kez140. PMID 31056705